CLINICAL TRIAL: NCT05258370
Title: "Exploration of the Role of Intact Fibroblast Growth Factor 23 and Its C-terminal Fragment in Chronic Respiratory Failure "
Brief Title: Fibroblast Growth Factor 23 in Chronic Respiratory Failure
Acronym: EFIC-RES
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Fondation Université de Paris (Unknown)
Responsible Party: Sponsor
Other Study IDs: APHP201305; 2020-A02607-32 (Other: ID-RCB Number - ANSM)
Record Dates: First submitted 2022-02-17; First posted 2022-02-28 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Chronic Respiratory Failure
Keywords: fibroblast growth factor 23; erythropoietin; cardiac hypertrophy; pulmonary hypertension; oxygen therapy; chronic respiratory failure
MeSH Terms: conditions — Cardiomegaly; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- incident patients with chronic respiratory failure: adult patients with untreated chronic respiratory failure
  Interventions: Other: Dosage; Other: Cardiac echography

INTERVENTIONS:
Other: Dosage — Evaluation of circulating C-terminal FGF23 (FGF23Ct) rate, circulating intact FGF23 (FGF23i) rate and Erythropoietin
Other: Cardiac echography — 12 months after patient enrollment

SUMMARY:
Fibroblast growth factor 23 (FGF23) is a key hormone of the mineral metabolism produced in bone and acting on the kidney to lower phosphatemia. FGF23 is subject to inactivating proteolytic cleavage which results in the presence of C-terminal and N-terminal fragments heretofore described as inactive.

We recently showed an increase in FGF23Ct in sickle cell patients, its association with left ventricular mass as well as a direct, pro-hypertrophic effect of FGF23Ct on rat cardiomyocytes. Data from the literature suggest that hypoxia (linked or not to anemia) is responsible for an increase in the production and cleavage of FGF23, either via the hypoxia inducible factor (HIF1α) or via the increase in erythropoietin (EPO).

We hypothesize that the FGF23Ct / FGF23i ratio is increased in response to chronic tissue hypoxia, in the absence of anemia, in patients with chronic respiratory failure (CRF) either due to a direct response to hypoxia via the stimulation of HIF1α, or indirectly via the increase in the circulating concentration of EPO. This elevation, if proven, could contribute to the increased risk of heart disease seen in some populations of CRF.

We propose to test this hypothesis by assaying FGF23Ct and FGF23i in a cohort of adult CRF patients before and after initiation of oxygen therapy.

The object of the present study is to study the FGF23Ct / FGF23i ratio in incident patients presenting with a non treated CRF as well as the modifications of this ratio under oxygen therapy and to study the correlations between FGF23 Ct and FGF23 and i) oxygen saturation and PaO2 ii) echocardiographic parameters and iii) EPO concentrations.

Three visits are planned: Baseline (before initiation of oxygen therapy), and two visits after initiation of oxygen therapy, at 3 months (M3) and at 12 months (M12).

For each visit, anthropometric and clinical data, treatment and biological results will be collected. FGF23 intact , FGF23 C-terminal and Erythropoietin will be measured. A cardiac ultrasound will be performed at baseline and at M12.

ELIGIBILITY:
Inclusion Criteria:

* Patient informed and not opposed to participating in the research
* Age ≥ 18 years old
* Severe chronic respiratory failure defined by PaO2 <60 mmHg, whatever the cause, and justifying the initiation of long-term oxygen therapy
* Not yet treated or with stopping oxygen therapy for at least 6 weeks
* Be affiliated with a social security scheme or be a beneficiary of such a scheme
* Be able to understand the interest and the constraints of the study

Exclusion Criteria:

* Exacerbation of respiratory failure in the 6 weeks prior to inclusion
* Chronic kidney disease defined by a glomerular filtration rate (GFR) estimated by CKD-EPI <60 mL / min / 1.73m2
* Anemia at the time of inclusion whatever the cause (sickle cell anemia, thalassemia, hemolytic anemia, chronic iron deficiency, others)
* Pregnancy
* Breastfeeding women
* Simultaneous participation in another therapeutic trial
* Patient under guardianship or curatorship
* Patient under medical help from the French government

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients with untreated chronic respiratory Ffilure with an indication to oxygen therapy and free from chronic kidney disease.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
circulating C-terminal FGF23 (FGF23Ct) | at inclusion (before oxygen therapy)
  ELISA method
circulating intact FGF23 (FGF23i) | at inclusion (before oxygen therapy)
  ELISA method

SECONDARY OUTCOMES:
circulating FGF23Ct | at month 3 and month 12
  ELISA method
circulating FGF23i | at month 3 and month 12
  ELISA method
circulating erythropoietin | at inclusion, month 3 and month 12
  ELISA method
arterial O2 saturation | at inclusion, month 3 (without and with 02 therapy) and month 12 (without and with 02 therapy)
  assessed using an arterial sampling
PaO2 (arterial partial oxygen pressure) | at inclusion, month 3 (without and with 02 therapy) and month 12 (without and with 02 therapy)
  assessed using an arterial sampling
Assessment of systolic function | at inclusion and month 12
  left ventricular ejection fraction assessed using cardiac ultrasound
left ventricular mass indexed for body surface area | at inclusion and month 12
  using cardiac ultrasound
Assessment of diastolic function | at inclusion and month 12
  Recording of mitral filling flow using cardiac ultrasound
Assessment of pulmonary artery pressure | at inclusion and month 12
  with measure, using cardiac ultrasound, of
  * The Vmax of the tricuspid insufficiency flow which gives the systolic gradient right heart ventricle/right heart atrium
  * And the diameter the inferior vena cava

CONTACTS AND LOCATIONS:
Overall Officials: Marie COURBEBAISSE, MD, Study Director — Assistance Publique - Hôpitaux de Paris; Nicolas ROCHE, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered.
  Data sharing must respect the agreements made with funders. Teams wishing obtain IPD must meet the sponsor and IP team to present scientific (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractual agreement.
  Processing of shared data must comply with European General Data Protection Regulation (GDPR).

REFERENCES:
- [Background] Courbebaisse M, Mehel H, Petit-Hoang C, Ribeil JA, Sabbah L, Tuloup-Minguez V, Bergerat D, Arlet JB, Stanislas A, Souberbielle JC, Le Clesiau H, Fischmeister R, Friedlander G, Prie D. Carboxy-terminal fragment of fibroblast growth factor 23 induces heart hypertrophy in sickle cell disease. Haematologica. 2017 Feb;102(2):e33-e35. doi: 10.3324/haematol.2016.150987. Epub 2016 Oct 27. No abstract available. PMID 27789679
- [Background] Clinkenbeard EL, Hanudel MR, Stayrook KR, Appaiah HN, Farrow EG, Cass TA, Summers LJ, Ip CS, Hum JM, Thomas JC, Ivan M, Richine BM, Chan RJ, Clemens TL, Schipani E, Sabbagh Y, Xu L, Srour EF, Alvarez MB, Kacena MA, Salusky IB, Ganz T, Nemeth E, White KE. Erythropoietin stimulates murine and human fibroblast growth factor-23, revealing novel roles for bone and bone marrow. Haematologica. 2017 Nov;102(11):e427-e430. doi: 10.3324/haematol.2017.167882. Epub 2017 Aug 17. No abstract available. PMID 28818868
- [Background] Zhang Q, Doucet M, Tomlinson RE, Han X, Quarles LD, Collins MT, Clemens TL. The hypoxia-inducible factor-1alpha activates ectopic production of fibroblast growth factor 23 in tumor-induced osteomalacia. Bone Res. 2016 Jul 5;4:16011. doi: 10.1038/boneres.2016.11. eCollection 2016. PMID 27468359
- [Background] Faul C, Amaral AP, Oskouei B, Hu MC, Sloan A, Isakova T, Gutierrez OM, Aguillon-Prada R, Lincoln J, Hare JM, Mundel P, Morales A, Scialla J, Fischer M, Soliman EZ, Chen J, Go AS, Rosas SE, Nessel L, Townsend RR, Feldman HI, St John Sutton M, Ojo A, Gadegbeku C, Di Marco GS, Reuter S, Kentrup D, Tiemann K, Brand M, Hill JA, Moe OW, Kuro-O M, Kusek JW, Keane MG, Wolf M. FGF23 induces left ventricular hypertrophy. J Clin Invest. 2011 Nov;121(11):4393-408. doi: 10.1172/JCI46122. Epub 2011 Oct 10. PMID 21985788